CLINICAL TRIAL: NCT03814967
Title: Transcranial Direct Current Stimulation (tDCS) Studies of Behavioral and Electrophysiological (EEG) Correlates of Higher-Order Cognition
Brief Title: Effects of Brain Stimulation on Higher-Order Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1344169; UCD#3565 (Other: University of CA Davis Psychiatry)
Record Dates: First submitted 2019-01-15; First posted 2019-01-24 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia
Keywords: schizophrenia; EEG; tDCS; dorsolateral prefrontal cortex; cognitive control; language; transcranial direct current stimulation
MeSH Terms: conditions — Schizophrenia; Language | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- DLPFC Stimulation (Experimental): Intervention. 20 minutes of 2 mA direct current stimulation over the dorsolateral prefrontal cortex.
  Interventions: Device: Transcranial Direct Current Stimulation
- Occipital Stimulation (Active Comparator): Intervention. 20 minutes of 2 mA direct current stimulation over the occipital cortex.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham Stimulation (Sham Comparator): Placebo Comparator. 0.5-1 minutes of 2 mA direct current stimulation over the dorsolateral prefrontal cortex followed by 19-19.5 minutes of sham stimulation
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — In tDCS, saline-soaked electrodes are temporary affixed to the scalp and connected to a battery-powered current generator. A weak (2 mA) constant current is then briefly applied (~20 minutes) to stimulate the targeted brain area (e.g. the DLPFC). To control for placebo effects, the study will utilize a sham stimulation protocol that consists of very brief constant stimulation (~1 minute). Subjects usually cannot discern the difference between the sham and experimental stimulation protocols due to habituation.

SUMMARY:
The purpose of this study is to better understand the neural correlates of higher-order cognition, both in the healthy brain and in schizophrenia, and to determine how these mechanisms are modulated by transcranial direct current stimulation (tDCS) at frontal and occipital scalp sites. Testing the effects of tDCS at these scalp sites on cognitive task performance will help us understand the roles of the brain regions corresponding to these sites during higher-order cognitive processing (language comprehension, cognitive control, and related attention and memory processes). Behavioral and electrophysiological (EEG) measures will be used to assess cognitive performance. The investigator's overarching hypothesis is that stimulating prefrontal circuits with tDCS can improve cognitive control performance, and ultimately performance on a range of cognitive tasks, as compared to stimulating a different cortical region (occipital cortex) or using sham stimulation. This study is solely intended as basic research in order to understand brain function in healthy individuals and individuals with schizophrenia. This study is not intended to diagnose, cure or treat schizophrenia or any other disease.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to sufficiently speak and understand English so as to be able to understand and complete cognitive tasks.
* All subjects must have the ability to give valid informed consent.

Inclusion Criteria for Patients with Schizophrenia Only:

* Diagnosis of schizophrenia, schizophreniform or schizoaffective disorder
* No medication changes in the prior month
* No medication changes anticipated in the upcoming month
* Stable outpatient or partial hospital status
* Normal IQ (>70; IQ will be measured by administering the Wechsler Abbreviated Scale of Intelligence (WASI) test)

Exclusion Criteria:

* Pacemakers
* Implanted electrical (brain and spinal) stimulators
* Implanted defibrillator
* Metallic implants
* Skin damage or skin conditions such as eczema at the sites where electrodes will be placed
* Hair styles hindering the placement of electrodes
* Cranial pathologies
* Head trauma
* Epilepsy
* Mental retardation
* Any known history of neurological disorders (including epilepsy, amyotrophic lateral sclerosis (ALS), multiple sclerosis (MS), stroke, cerebral palsy, any DSM-5 axis I psychiatric disorder (for healthy control subjects), autism)
* Uncorrected vision problems that would hinder cognitive testing (this also pertains to subjects with color blindness in tasks where discriminating colored objects/items is necessary for successful performance)
* Pregnancy
* Substance dependence in the past six months
* Substance abuse in the past month

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
EEG Correlates of Language and Cognitive Control | Assessment will begin immediately following stimulation and last for about 1.5 hours.
  Electrophysiological data recorded during completion of cognitive control and language comprehension tasks. We will measure oscillatory activity in the theta, alpha, beta and gamma frequency bands.
Behavioral Response (Cognitive Control Task) | Assessment will begin immediately following stimulation and last for about 1.5 hours.
  We will assess performance on the Dot Pattern Expectancy (DPX) task (error rates and d-prime scores).
Behavioral Response (Language Task) | Assessment will begin immediately following stimulation and last for about 1.5 hours.
  We will assess performance on a novel Language Comprehension task (accuracy and semantic relatedness judgement scores).

CONTACTS AND LOCATIONS:
Locations (1):
- Imaging Research Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Select data from this study may be submitted to the National Institute of Mental Health Data Archive (NDA). NDA is a data repository run by the National Institute of Mental Health (NIMH) that allows researchers studying mental illness to collect and share de-identified information with each other. The data repository is accessible only to qualified investigators. All subject data will be de-identified (subject names will not be used) and each subject will have a separate identifier called a Global Unique Identifier (GUID) to remove any possibility that "the identities of the subjects cannot be readily ascertained or otherwise associated with the data by the repository staff or secondary data users." (45 CFR, 46.102).

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-study-of-the-effects-of-brain-stimulation-on-higher-order-cognition-761403/